CLINICAL TRIAL: NCT04730401
Title: Randomized, Double-Blind, Placebo-Controlled Study of Convalescent Plasma in the Treatment of Covid-19
Brief Title: Convalescent Plasma in the Treatment of Covid-19
Acronym: CP_COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Finnish Red Cross Blood Service (Other)
Responsible Party: Principal Investigator, Anu Kantele, Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Plasma_Covid-19
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Covid19
Keywords: Covid-19; Convalescent plasma; Safety
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Some of the investigators are masked and some are not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-titre CP (Experimental): 200mL high-titre CP on admittance
  Interventions: Biological: Convalescent plasma from COVID-19 donors
- low-titre CP (Active Comparator): 200ml low-titre CP on admittance
  Interventions: Biological: Convalescent plasma from COVID-19 donors
- Placebo (Placebo Comparator): 200mL saline as placebo on admittance
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Convalescent plasma from COVID-19 donors — Convalescent plasma from COVID-19 donors
  Arms: High-titre CP; low-titre CP
Biological: Placebo — 200mL saline
  Arms: Placebo

SUMMARY:
This study investigates the possible adverse effects and effectiveness of convalescent plasma for patients infected with SARS-CoV-2. Following provision of informed consent, patients will be randomized into three groups: High-titre convalescent plasma, low-titre convalescent plasma or placebo. Primary outcomes of the study will cover safety and either intubation or initiation of systemic corticosteroids. Safety information collected will include serious adverse events judged to be related to administration of convalescent plasma. Microbiological and other laboratory parameters will be followed up.

DETAILED DESCRIPTION:
SARS-CoV-2 pandemic presents a serious global public health threat urgently requiring both prophylactic and therapeutic interventions. The entry of SARS-CoV-2 into human cells involves a binding between its spike protein's receptor-binding domain (RBD) and angiotensin-converting enzyme 2 (ACE2) receptor on human cells. Convalescent sera of Covid-19 patients have been shown to contain SARS-CoV-2-neutralizing antibodies. Accordingly, recovered patients are presumed to be immune to re-infection. Use of convalescent plasma as treatment warrants research, which is supported by the European Commission. Convalescent plasma (CP) therapy is a classical adaptive immunotherapy. It has been applied to prevention and treatment of various infectious diseases: evidence of success has been accumulated e.g. on treatment of SARS, MERS, and 2009 H1N1, for which satisfactory efficacy and safety have been shown.

The investigators will select as donors for CP therapy patients recovered from Covid-19 with a high neutralizing antibody titre who meet normal blood donor eligibility criteria. The donors will be recruited among participants of ongoing Covid-19 immunity studies (Clin-Covid, Commun-Covid) and/or from Finnish Red Cross Blood Service (FRCBS) blood donors.

CP will be prepared from the blood of eligible donors at the FRCBS according to previous protocols and the European guidelines for fresh frozen plasma. After the screening test results required for product release (HCV, HBV, HIV, ABO, Syphilis) are available, the units will be released. All donors will be screened for type-I-Interferon antibodies and women will be screened for HLA-antibodies. The units will be labelled with convalescence plasma labels including ICCBBA/ISBT compliant product codes. The plasma units will be frozen to -25°C within 6 hours from collection. Prior to freezing 3 ml of CP will be separated and divided in 3 aliquots to be stored, for possible later analysis.

Patients admitted to ward at HUH will be randomized 1:1:1 into three groups which will be given 1) high-titre convalescent plasma (HCP), 2) low-titre convalescent plasma (LCP) or 3) placebo. The plasma preparations and placebo will be given as one 200 mL infusion. ABORh blood group will be determined from patients prior to transfusion according to normal transfusion protocols of the hospital. The study will be double-blinded with saline as placebo given to groups three. The primary outcomes of the study will cover safety and intubation/initiation of systemic corticosteroids. AEs will be reviewed, recorded and reported up to 6 hours after administration of CP or placebo. Thromboembolic and cardiovascular events will be recorded as AEs or SAEs up to 7 days after administration of CP / placebo. SAEs will be reviewed, recorded and reported up to 7 days after administration of CP / placebo. In case of respiratory failures classified as SAEs, the reporting period is only up to 12 hours after administration of CP / placebo.

ELIGIBILITY:
Inclusion Criteria:

* Acute Covid-19 disease at the time of recruitment laboratory-confirmed by upper respiratory tract PCR
* Patient recently (0-4 days earlier) admitted to hospital due to Covid-19 infection
* Symptom onset 10 days before recruitment (if symptom onset unknown the duration is calculated from positive PCR-test)
* the day should be recorded from the duration of the Covid-19 symptoms/positive test result
* The dose of LMWH thromboprofylaxis should be recorded
* Written informed consent.

Exclusion Criteria:

* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of IMP; oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent are excluded ( inhaled or topical steroids allowed)
* Regular (daily), systemic administration of corticosteroids at the time on inclusion (inhaled or topical corticosteroids are allowed)
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Pregnancy or lactation.
* Alcohol or drug abuse.
* Suspected non-compliance.
* Presence of VTE, including pulmonary embolism or other manifestations of thrombosis
* Use of any investigational drug (other than hydroxychloroquine) or vaccine within 30 days prior to first dose of study vaccine or planned use during study period.
* Any clinically significant history of known or suspected anaphylaxis or hypersensitivity reaction as judged by investigator.
* Known immunoglobulin A (IgA) deficiency
* Existing treatment limitations: do-not-resuscitate (DNR) order or withholding treatment in ICU
* Any other criteria which, as judged by investigator, might compromise a patient's well-being or ability to participate in the study or its outcome.
* Active malignant disease
* CP not available for patients blood type
* Patient cannot assign written consent
* No personnel available for CP of placebo transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety (SAE) | SAEs will be reviewed, recorded and reported up to 6 hours after administration of CP or placebo.
  Immediate serious adverse events (SAE) between active and non-active group
Safety (SAE) | SAEs will be recorded and reported up to 7 days after administration of CP or placebo.
  Subsequent serious adverse events (SAE) between active and non-active group
Rate of intubation or systemic corticosteroids initiation | 21 days post transfusion
  Intubation or systemic corticosteroid treatment (e.g. dexamethasone) started for aggravation of Covid-19

SECONDARY OUTCOMES:
Hospital stay | Through study completion, up to 1 year
  Number of days at hospital during the COVID-19 infection hospital period
Mortality | Through study completion, up to 1 year
  Proportion of fatal cases during the COVID-19 infection hospital period
Mortality | 21 days post transfusion
  Proportion of fatal cases during the COVID-19 infection hospital period
ICU stay | Within 21 days post transfusion
  Number of ICU days during the COVID-19 infection hospital period
Ventilator days | Within 21 days post transfusion
  Number of ventilator days during the COVID-19 infection hospital period
Severity of respiratory failure | 21 days post transfusion
  Highest severity of respiratory failure using adapted WHO Clinical Progression Scale
Viral load | During hospitalizaation, through study completion, up to 1 year
  Analyses of respiratory tract secretions by SARS-CoV-2 PCR during the COVID-19 infection hospital period
Antibody measurements | Through study completion, up to 1 year
  Analyses of SARS-CoV-2-specific antibodies in serum and excretions
Thrombotic complication | Through study completion, up to 1 year
  Development of a thrombotic complication, including VTE or arterial thrombosis
The rate of participants presenting with coagulopathy disorders | 21 days post transfusion
  Development of sepsis-induced coagulopathy or disseminated intravascular coagulation during the COVID-19 infection hospital period
Number of participants with laboratory change | Through study completion, up to 1 year
  Change in inflammatory (CRP, Ferritin) and coagulopathy (P -APTT, P -AT3, P -Fibr, P -FiDD, P -FVIII., P -Trombai ja P -TT) markers during the COVID-19 infection hospital period
Adverse effects | Through study completion, up to 1 year
  Comparison of adverse events between active and non-active group
Convalescent plasma efficacy | 21 day post transfusion
  Convalescent plasma (high or low titer) efficacy versus placebo: rate of intubation or initiating systemic corticosteroids during the COVID-19 infection hospital period
Convalescent plasma high vs low titer efficacy | 21 day post transfusion
  Comparison of efficacy of high titer CP to low titer CP: Rate of intubation or initiating systemic corticosteroids during the COVID-19 infection hospital period
Convalescent plasma efficacy according to donor status | 21 day post transfusion
  Comparison of efficacy CP obtained from vaccinated donors versus non-vaccinated donors: Rate of intubation or initiating systemic corticosteroids during the COVID-19 infection hospital period

CONTACTS AND LOCATIONS:
Overall Officials: Anu Kantele, MD,Prof, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No